CLINICAL TRIAL: NCT04748913
Title: Diagnostic Accuracy of Near Infrared Transillumination in Combination With a Dye in the Cavitation Detection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad Rey Juan Carlos (Other)
Responsible Party: Principal Investigator, Santiago Miguel de Vega Calleja, Principal investigator, Universidad Rey Juan Carlos
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: Universidad Rey Juan Carlos
Record Dates: First submitted 2021-02-02; First posted 2021-02-10 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Initial Proximal Caries
MeSH Terms: interventions — Diagnostic Imaging; Radionuclide Imaging

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No intervention (No Intervention)
- Remineralization (Other)
  Interventions: Device: Radiographic examination; Device: Scanning with DIAGNOcam; Device: Scan with DIAGNOcam and Indocyanine; Diagnostic Test: Visual-tactile exploration with separation

INTERVENTIONS:
Device: Radiographic examination — Standardized bitewing radiographs will be performed by the principal investigator
  Arms: Remineralization
Device: Scanning with DIAGNOcam — The surface of the selected teeth will be examined under near infrared light using the DIAGNOcam device
  Arms: Remineralization
Device: Scan with DIAGNOcam and Indocyanine — One the dye has been applied, a new series of images will be taken with Diagnocam
  Arms: Remineralization
Diagnostic Test: Visual-tactile exploration with separation — The point of contact will be open in the corresponding proximal area of the lesion using an elastic orthodontic separator
  Arms: Remineralization

SUMMARY:
The aim of the study will be to make a comparison in vivo of the following techniques:

DIAGNOcam, DIAGNOcam in combination with indocyanine and bitewing radiography, analyzing the ability to detect cavitation in initial proximal caries in posterior teeth using visual separation with tactile exploration as a gold standard.

Methodology:

During a period of 2 years, patients with initial proximal caries will be evaluated in the facilities of the clinic belonging to the Fundación de la Clínica Universitaria of the Rey Juan Carlos University (Madrid, Spain). Those subjects where a minimum of a proximal carious lesion (E1, E2 or D1) is diagnosed in posterior teeth will be candidates for the study. The exploration of proximal caries will be carried out in four phases: radiographic exploration, exploration with DIAGNOcam, exploration with DIAGNOcam and Indocyanine and visual-tactile exploration with separation. Once the visual-tactile examination with separation has been completed, the caries lesions will be treated. Depending on whether the lesion is cavitated or not, a non-invasive procedure or an operative treatment will be chosen.

ELIGIBILITY:
Inclusion Criteria:

* E1, E2 and D1 proximal carious lesions in permanent posterior teeth (E1: outer half of enamel; E2: inner half of enamel; D1: outer half of dentin)

Exclusion Criteria:

* estructural abnormalities
* visible clinical cavitation
* restorations on the proximal surfaces
* open contact points
* overlapping structures on the X-ray that prevent a clear view of the proximal area

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-11-09 (Actual); Primary Completion 2022-11-09 (Estimated); Study Completion 2022-11-09 (Estimated)

PRIMARY OUTCOMES:
Near infrared transillumination | 2 years
  Ability to detect cavitation in initial proximal caries of DIAGNOcam in combination with indocyanine

CONTACTS AND LOCATIONS:
Locations (1):
- Santiago De Vega Calleja, Alcorcón, Madrid, Spain